CLINICAL TRIAL: NCT04786132
Title: The Effects of 8-week Cognitive-motor Training on Proprioception and Postural Control Under Single and Dual Task Conditions in Healthy Older Adults: A Randomized Clinical Trials.
Brief Title: The Effects of Cognitive-motor Training in Healthy Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Ramon Llull (Other)
Collaborators: Ainhoa Nieto Guisado (Unknown); Mónica Solana-Tramunt (Unknown)
Responsible Party: Principal Investigator, Jose Morales, Principal investigator, University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0.2 Dual task
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Proprioception Change; Balance Change; Cognitive Change
Keywords: Dual Task; Proprioception; Balance; Music

STUDY DESIGN:
Intervention Model Description: Pre test, intervention and Post test. Experimental group performs and eight week dual task training with proprioception and balance exercise while including unknown sung music 2 days a week. Control group do the same protocol and the same days but without the inclusion of music.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task (proprioception, balance and cognitive) training (Experimental): A DT training protocol of 8 weeks duration was carried out, during 2 days a week, with a duration of 30 minutes each session divided into: warm-up (mobility and warm-up 5 '), main part (20') and cool down (5 'dynamic stretching). The main part consisted of a choreography divided into five measures of thirty-two beats each, in turn divided into four parts of eight movements, which included proprioception and balance exercises such as: squats, imbalances, lateral movements, front, standing on one leg, twist, etc. The sessions evolved from individual exercises, in pairs, in trios and finally in groups. The sessions included music that was unknown to the subjects but at the same time easy to learn, so that while they performed the motor tasks, they would memorize the songs.
  The sessions were carried out by the main researcher who controlled both the technique of the exercises and motivated them to sing and perform a cognitive exercise.
  Interventions: Other: Cognitive-motor training
- Proprioception and balance training (Active Comparator): The control group training protocol is the same as the experimental group, whit the same duration and the same sessions, the unique difference is that there was no music included in the sessions, and therefore cognitive ability was not worked.
  The sessions were carried out by the main researcher who controlled the technique of the exercises and motivated the participant.
  Interventions: Other: Motor training

INTERVENTIONS:
Other: Cognitive-motor training — A DT training protocol of 8 weeks duration was carried out, during 2 days a week, with a duration of 30 minutes each session divided into: warm-up (mobility and warm-up 5 '), main part (20') and cool down (5 'dynamic stretching). The main part consisted of a choreography divided into five measures of thirty-two beats each, in turn divided into four parts of eight movements, which included proprioception and balance exercises such as: squats, imbalances, lateral movements, front, standing on one leg, twist, etc. The sessions evolved from individual exercises, in pairs, in trios and finally in groups. The sessions included music that was unknown to the subjects but at the same time easy to learn, so that while they performed the motor tasks, they would memorize the songs.
  The sessions were carried out by the main researcher who controlled both the technique of the exercises and motivated them to sing and perform a cognitive exercise.
  Arms: Dual Task (proprioception, balance and cognitive) training
Other: Motor training — A training protocol of 8 weeks duration was carried out, during 2 days a week, with a duration of 30 minutes each session divided into: warm-up (mobility and warm-up 5 '), main part (20') and cool down (5 'dynamic stretching). The main part consisted of a choreography divided into five measures of thirty-two beats each, in turn divided into four parts of eight movements, which included proprioception and balance exercises such as: squats, imbalances, lateral movements, front, standing on one leg, twist, etc. The sessions evolved from individual exercises, in pairs, in trios and finally in groups.
  Arms: Proprioception and balance training

SUMMARY:
Currently, there is a growing concern for the elderly population and for what the increase in life expectancy entails, and that is why many authors investigate about exercise protocols that delay the appearance of both cognitive and motor diseases and how to link both in your day to day. Despite this, there is still little information about training with DT tasks that improve the life of the elderly and that is why this study aims to evaluate the effect of an eight-week training program in older adults healthy, in the improvement of balance and proprioception of the knee, with the inclusion of a cognitive task performed simultaneously. We hypothesize that the inclusion of the double motor-cognitive task in the training sessions will improve the performance in the balance and proprioception tests performed with the simultaneous cognitive task after 8 weeks compared to the control group.

DETAILED DESCRIPTION:
The study included the participation of 30 physically active older adults, who were recruited in a sports center in the community of Cataluña, between the ages of 65-85 years. Potential participants were excluded from the sample if they: i) suffered from a neurological condition such as Alzheimer's or Parkinson's disease ii) were unable to perform one or more of the parts of testing and/or iii) were undergoing pharmacological treatments likely to alter postural control and proprioception, iv) underwent lower limb joint replacement surgery. The participants were invited to take part in the study voluntarily and they were informed verbally and in writing as to the characteristics of the programme.

The study was carried out in accordance with the ethical standards set out according to the Declaration of Helsinki, and it was approved by the Ethics Committee at Ramón Llull University. All protocols applied in this research (including the management of the personal data of the participants) complied with the requirements specified in the Declaration of Helsinki of 1975 and its subsequent revisions.

The specific DT program is aimed at physically active people between 8 and 15 years old who train at the center in maintenance classes for the elderly and aim to improve their quality of life and keep them active for the functionality of their daily lives. All the study participants will be asked to sign an informed consent document that will be drafted in keeping with all applicable research ethics protocols, including a guarantee of the confidentiality of personal data and an assurance that participants can choose to abandon the study at any time.

Control group (CG), experimental group (EG) and pre-test, post-test methodology was selected. EG performed the specific DT while CG carried out the motor training.

The motor-cognitive intervention will be carried out over one year in the years (2019-2020). The first 3 months allowed investigators to recruit the participants and and observe the training sessions that the subjects did in the center. After this, the researchers designed an intervention that complemented the training that the subjects had previously carried out and were specific training for the study objectives.

This design took into account the previous experiences of the subjects' trainer and of an expert physical therapist in motor control (balance and proprioception), and a psychologist. Before starting the real intervention, test sessions of the training protocol to be developed were applied to know the level of the subjects, and thus have data that would allow us to adjust the training schedule to their needs and abilities. The conclusions drawn from this initial experience formed the scientific basis for the definitive version of motor-cognitive training.

During the fourth month, a preliminary test was carried out that included 4 balance tests, a propioceptive test and a cognitive test. The participants performed the tests in an isolated, comfortable place that did not interfere with their results. The order of the subjects and the order of the applied tests were determined randomly using a true random number generator to avoid order effects. An expert team of researchers in the field directed and controlled the tests.

Romberg test: it was the test selected to measure the motor control of the participants. Three measurement conditions were used: bipedal eyes open / eyes closed and unipedal dominant eyes open. Balance was measured on a KISTLER force platform.

Proprioception: To evaluate proprioception, the absolute repositioning error of the knee joint at 45 degrees (AEr45º) in the dominant leg was recorded. This measurement was taken with the Goniometer Pro mobile application.

Subscale of the Barcelona Test: to carry out the performance of the dual task, the subjects performed a cognitive task while their balance and proprioception were evaluated. The cognitive task came from the subscale called "categorical evocation in associations", which is found within the battery of subscales of the Revised Barcelona Test. The task consisted of mentioning the maximum number of possible words for 30 seconds belonging to the same semantic field.

In all this tests, the participants wore an orthopedic boots on both feet for the postural control measurements, helping to guarantee that the two tests (postural control and proprioception) would yield comparable results. These boots served to eliminate the effects of any initial postural control adaptations made by the toes or ankle, thus ensuring that the knee would act as the main balancing mechanism.

From October to December, the cognitive-motor training sessions were carried out in the same room in which the participants previously carried out their activities, and at the same time, thus guaranteeing the safety of the participants. An instructor will lead the session and the monitor of the activities of the participants will reinforce and help during the exercise protocol. Two sessions were held per week, on different days for each of the groups, in order not to create interferences or learning in the subjects. The duration of the sessions was thirty minutes and it was divided into a five-minute warm-up, the main part of twenty minutes and a cool down of five minutes. During the main part it was controlled that the technical execution of the exercises was carried out correctly in order to avoid injuries and favor the improvement of the balance and proprioception of the participants.

The main part consisted of a simple choreography, which progressed in the difficulty of the exercises after the sessions. It began with individual balance and proprioception exercises in the first session, in pairs in the second, trios for the third, and in groups of four for the fourth, and until the end of the protocol. The proposed exercises included walking, lateral movements, forward and backward, simple balances with both legs, and more complex when performed in the company of others, knee bends at no more than 45º to be related to the proprioception tests. For example, when performing a squat, imbalances were proposed with pairs or trios to compromise the stability of the participants, or dances such as the twist or the conga to, in addition to working on balance, promoted socialization and fun for the participants. The only difference in the training protocol between CG and EG was the inclusion of sung music in EG sessions. The objective was that at the end of the 4 sessions listening to the same music, the subjects learned pieces of the songs and that during the training they were singing them or at least memorizing them.

A post-test was carried out once the 8 weeks of the intervention protocol had ended, as was the pre-test protocol.

The Statistical Analysis will be executed using an Excel sheet and then it will be exported to the SPSS Statistics 22.0 computer program, to then carry out the different statistical tests. Initially, a normality test will be run to verify the distribution of the data and decide whether to apply parametric or nonparametric tests. The G-POWER program will be used to calculate the statistical power of the sample with a value of p <0.05 and an estimated effect size of 0.5.

ELIGIBILITY:
Inclusion Criteria:

* Physically active older adults

Exclusion Criteria:

* Clinical disability for physical activity
* Neurological condition such as Alzheimer's or Parkinson's disease
* Subjected to drug treatments that alter the normal functioning of the nervous system
* Recent lower limb joint replacement surgery (12 months before testing)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Motor control results | Up to 8 weeks
  Change from pre-test to post-test in motor control results. The bipedal and unipodal Romberg Test was performed to evaluate the balance of the subjects. Variants of open and closed eyes were applied for the bipedal test and dominance for the unipedal test, in order to find more difference between groups. These tests were performed on a force platform, considered a gold standard tool for the analysis of postural balance deficits, using valid parameters and confidence stabilometry measures. The recorded values were the area of the ellipse and the mean velocity in the anterior-posterior (MVAP) and medial-lateral (MVML) directions. While the area of the ellipse acts as an indicator of postural control performance, MVAP and MVML readings provide information on the neuromuscular activity used to maintain postural control (Frederic Noé & Paillard, 2005). For all these variables, lower scores indicate better performance on tasks.
Proprioception results | Up to 8 weeks
  Change from pre-test to post-test in proprioception results. The AEr45º in the dominant leg was recorded. This measurement was taken using the Goniometer Pro mobile app (2.9, 5Fuf5 co, Bloomfield, NJ, United States). It provides instantaneous, accurate, repeatable readings of the range of movement (ROM), measuring the difference between the required knee angle and the position that is observed (Mourcou et al., 2016). During the test, participant close their eyes, placed their knees at a 45º angle and maintain this position for six seconds and return to the original standing position. Afterwards they were told to bend their knees again until they had returned to exactly the same position the researcher had placed them in (i.e. 45º). In order to quantify conscious proprioception the absolute value of the difference between the requested (45º) and the actual angle was recorded to determine the participant's joint repositioning ability.
Cognitive results | Up to 8 weeks
  Change from pre-test to post-test in cognitive results The cognitive task came from the subscale called "categorical evocation in associations", which is found within the battery of subscales of the Revised Barcelona Test (Peña-Casanova, 2005). The task consisted of mentioning the maximum number of possible words for 30 seconds belonging to the same semantic field. The semantic fields chosen were the following: 1. Animals; 2.Fruit; 3. Cities; 4. Parts of the body; 5. Garments; 6.Meals; 7. Countries; 8.Colors; 9. Names of women; 10. Names of men. The score obtained depends on the number of words remembered, scoring a point for each of them. No points were added to repeated words or synonyms (Peña-Casanova, 2005). To quantify the total number of words that the subjects said, they were recorded and once the tests were finished, the total of words mentioned in each repetition were counted.

SECONDARY OUTCOMES:
Cognitive Reserve Results | Only measured at the beginning of the intervention
  To know the cognitive reserve of the subjects, they answered a validated questionnaire of the CR scale, which consisted of 24 questions related to their lifestyle (studies, hobbies, physical activity, reading, music, languages, etc.) (León et al., 2014). They had to answer how often in their Youth, Adulthood, and Maturity (currently), they performed such activities with the following response code: following response code: 0 = Never; 1 = Once or several times a year; 2 = Once or several times a month; 3 = Once or several times a week; 4 = Three or more times a week, whenever the opportunity arises. Once concluded, the scores were added and the higher the better the cognitive reserve, which translates into a higher educational and occupational level throughout their life, a better cognitive reserve, benefiting this to better brain function (Rodríguez Álvarez & Sánchez Rodríguez , 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Solana-Tramunt, Study Director — University Ramon Llull
Locations (1):
- Ainhoa Nieto Guisado, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stern Y. Cognitive reserve. Neuropsychologia. 2009 Aug;47(10):2015-28. doi: 10.1016/j.neuropsychologia.2009.03.004. Epub 2009 Mar 13. PMID 19467352
- [Background] Wang H, Ji Z, Jiang G, Liu W, Jiao X. Correlation among proprioception, muscle strength, and balance. J Phys Ther Sci. 2016 Dec;28(12):3468-3472. doi: 10.1589/jpts.28.3468. Epub 2016 Dec 27. PMID 28174475
- [Background] Liu Y, Lachman ME. Education and Cognition in Middle Age and Later Life: The Mediating Role of Physical and Cognitive Activity. J Gerontol B Psychol Sci Soc Sci. 2020 Aug 13;75(7):e93-e104. doi: 10.1093/geronb/gbz020. PMID 30955036
- [Background] Kim SJ, Yoo GE. Rhythm-Motor Dual Task Intervention for Fall Prevention in Healthy Older Adults. Front Psychol. 2020 Jan 17;10:3027. doi: 10.3389/fpsyg.2019.03027. eCollection 2019. PMID 32010035
- [Background] Hiyamizu M, Morioka S, Shomoto K, Shimada T. Effects of dual task balance training on dual task performance in elderly people: a randomized controlled trial. Clin Rehabil. 2012 Jan;26(1):58-67. doi: 10.1177/0269215510394222. Epub 2011 Mar 18. PMID 21421689